CLINICAL TRIAL: NCT01960686
Title: A Phase II Randomized, Observer-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Immunogenicity and Safety of Multiple Formulations of an RSV F Particle Vaccine With Aluminum, in Healthy Women of Child-Bearing Age
Brief Title: RSV F Dose-Ranging Study in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NVX757.M202
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Low dose RSV F Vaccine with Dose 1 of Aluminum Adjuvant (Experimental): Day 0: Low dose RSV F Antigen with Dose 1 of aluminum adjuvant Day 28: Placebo
  Interventions: Biological: Low dose RSV F Antigen; Biological: Dose 1 of Aluminum Adjuvant; Biological: Placebo
- Low dose RSV F Vaccine with Dose 2 of Aluminum Adjuvant (Experimental): Day 0: Low dose RSV F Antigen content with Dose 2 of aluminum adjuvant Day 28: Low dose RSV F Antigen content with Dose 2 of aluminum adjuvant
  Interventions: Biological: Low dose RSV F Antigen; Biological: Dose 2 of Aluminum Adjuvant
- Low dose RSV F Vaccine with Dose 3 of Aluminum Adjuvant (Experimental): Day 0: Low dose RSV F Antigen with Dose 3 of aluminum adjuvant Day 28: Low dose RSV F Antigen with Dose 3 of aluminum adjuvant
  Interventions: Biological: Low dose RSV F Antigen; Biological: Dose 3 of Aluminum Adjuvant
- Low dose RSV F Vaccine with Dose 4 of Aluminum Adjuvant (Experimental): Day 0: Low dose RSV F Antigen with Dose 4 of aluminum adjuvant Day 28: Low dose RSV F Antigen with Dose 4 of aluminum adjuvant
  Interventions: Biological: Low dose RSV F Antigen; Biological: Dose 4 of Aluminum Adjuvant
- High dose RSV F Vaccine with Dose 2 of Aluminum Adjuvant (Experimental): Day 0: High dose RSV F Antigen with Dose 2 of aluminum adjuvant Day 28: Placebo
  Interventions: Biological: High dose RSV F Antigen; Biological: Dose 2 of Aluminum Adjuvant; Biological: Placebo
- High dose RSV F Vaccine with Dose 3 of Aluminum Adjuvant (Experimental): Day 0: High dose RSV F Antigen with Dose 3 of aluminum adjuvant Day 28: Placebo
  Interventions: Biological: High dose RSV F Antigen; Biological: Dose 3 of Aluminum Adjuvant; Biological: Placebo
- High dose RSV F Vaccine with Dose 4 of Aluminum Adjuvant (Experimental): Day 0: High dose RSV F Antigen content with Dose 4 of aluminum adjuvant Day 28: Placebo
  Interventions: Biological: High dose RSV F Antigen; Biological: Dose 4 of Aluminum Adjuvant; Biological: Placebo
- Placebo (Placebo Comparator): Day 0: Placebo Day 28: Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dose RSV F Antigen
  Arms: Low dose RSV F Vaccine with Dose 1 of Aluminum Adjuvant; Low dose RSV F Vaccine with Dose 2 of Aluminum Adjuvant; Low dose RSV F Vaccine with Dose 3 of Aluminum Adjuvant; Low dose RSV F Vaccine with Dose 4 of Aluminum Adjuvant
Biological: High dose RSV F Antigen
  Arms: High dose RSV F Vaccine with Dose 2 of Aluminum Adjuvant; High dose RSV F Vaccine with Dose 3 of Aluminum Adjuvant; High dose RSV F Vaccine with Dose 4 of Aluminum Adjuvant
Biological: Dose 1 of Aluminum Adjuvant
  Arms: Low dose RSV F Vaccine with Dose 1 of Aluminum Adjuvant
Biological: Dose 2 of Aluminum Adjuvant
  Arms: High dose RSV F Vaccine with Dose 2 of Aluminum Adjuvant; Low dose RSV F Vaccine with Dose 2 of Aluminum Adjuvant
Biological: Dose 3 of Aluminum Adjuvant
  Arms: High dose RSV F Vaccine with Dose 3 of Aluminum Adjuvant; Low dose RSV F Vaccine with Dose 3 of Aluminum Adjuvant
Biological: Dose 4 of Aluminum Adjuvant
  Arms: High dose RSV F Vaccine with Dose 4 of Aluminum Adjuvant; Low dose RSV F Vaccine with Dose 4 of Aluminum Adjuvant
Biological: Placebo
  Arms: High dose RSV F Vaccine with Dose 2 of Aluminum Adjuvant; High dose RSV F Vaccine with Dose 3 of Aluminum Adjuvant; High dose RSV F Vaccine with Dose 4 of Aluminum Adjuvant; Low dose RSV F Vaccine with Dose 1 of Aluminum Adjuvant; Placebo

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of multiple formulations of an RSV-F protein nanoparticle vaccine, with aluminum, in healthy women of child-bearing age.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be eligible to participate:

1. Healthy adult females, ≥ 18 and ≤ 35 years of age. "Healthy" shall be defined by the absence of any illness, acute or chronic, that requires ongoing systemic therapy for the control of symptoms or prevention of disability.

   * Subjects on stable (no change in ≥ 3 months) therapy for findings (e.g., hypertension or hyperlipidemia) that are not associated with symptoms or disability are eligible, as are users of hormonal contraceptives.
   * Subjects who receive intermittent prophylaxis for risks associated with asymptomatic findings (e.g., antibiotic prophylaxis prior to dental procedures in a subject with mitral valve prolapse) are eligible.
   * Ongoing therapy will be defined as continuous or, if intermittent, more frequent than once every 3 months (e.g., use of an inhaled bronchodilator for exercise-induced bronchospasm more than once every 3 months). Immunosuppressives are subject to exclusion criterion #5 below.
   * Persons being treated for illnesses or conditions that would become acutely symptomatic or disabling in the absence of treatment are not eligible.
2. Willing and able to give informed consent prior to study enrollment.
3. Able to comply with study requirements.
4. Women who are not surgically sterile must have a negative urine pregnancy test prior to each vaccination; will be advised through the Informed Consent process to avoid becoming pregnant over the duration of the study, and must assert that they will employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: credible history of continuous abstinence from heterosexual activity, hormonal contraceptives (oral, injectable, implant, patch, ring), double-barrier contraceptives (condom or diaphragm, with spermicide), and IUD.

Exclusion Criteria:

Subjects will be excluded if they fulfill any of the following criteria:

1. Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of first vaccination.
2. History of a serious reaction to any prior vaccination.
3. Received any vaccine in the 4 weeks preceding the study vaccination; or any RSV vaccine at any time.
4. Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
5. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
6. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
7. Donated blood within 3 weeks of the planned date of first vaccination.
8. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C on the planned day of vaccine administration).
9. Known disturbance of coagulation.
10. Women who are pregnant or breastfeeding, or plan to become pregnant during the study.
11. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.
12. Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 720 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Immunogenicity as assessed by serum IgG antibody titers specific for the F-Protein antigen across treatment groups | Day 0 to Day 56
  Serum IgG antibody concentrations as ELISA units (EUs) specific for the F protein antigen.
  Derived/calculated endpoints based on these data will include:
  * Geometric mean concentrations as EU (GMEU)
  * Geometric mean ratio (GMR)
  * Geometric mean fold-rise (GMFR)
  * Seroconversion rate (SCR)
  * Seroresponse rate (SRR)
Assessment of Safety | Day 0 to Day 182
  Numbers and percentages of subjects with solicited local and systemic adverse events over the seven days post-injection; and all adverse events, solicited and unsolicited, including adverse changes in clinical laboratory parameters. In addition, Medically Attended Events, Serious Adverse Events, and Significant New Medical Conditions will be collected for six months.

SECONDARY OUTCOMES:
Immunogenicity based on neutralizing antibody titer | Day 0 to Day 56
Kinetics of serum IgG antibody titers specific for the F-Protein antigen across time | Day 0 to Day 91
Immunogenicity based on antibodies sharing specificity with Palivizumab | Day 0 to 91

CONTACTS AND LOCATIONS:
Overall Officials: D. Nigel Thomas, Ph.D., Study Director — Novavax, Inc.
Locations (10):
- United States (10):
  - Diablo Clinical Research, Walnut Creek, California
  - Clincal Research of Atlanta, Stockbridge, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Johnson County Clin-Trials, Lenexa, Kansas
  - QPS Bio-Kinetic, Springfield, Missouri
  - Wake Research Associates, Raleigh, North Carolina
  - Coastal Carolina Research, Mt. Pleasant, South Carolina
  - Research Across America, Dallas, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Derived] August A, Glenn GM, Kpamegan E, Hickman SP, Jani D, Lu H, Thomas DN, Wen J, Piedra PA, Fries LF. A Phase 2 randomized, observer-blind, placebo-controlled, dose-ranging trial of aluminum-adjuvanted respiratory syncytial virus F particle vaccine formulations in healthy women of childbearing age. Vaccine. 2017 Jun 27;35(30):3749-3759. doi: 10.1016/j.vaccine.2017.05.045. Epub 2017 Jun 1. PMID 28579233